CLINICAL TRIAL: NCT01876030
Title: Comparison of Different Treatment Methods for Gait Rehabilitation of Sub-Acute Post Stroke Patients With Dropped Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyGait-HMO-CTIL
Record Dates: First submitted 2013-05-02; First posted 2013-06-12 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Dropped Foot
Keywords: Functional electrical stimulation (FES); Sub acute stroke; Gait analysis
MeSH Terms: conditions — Peroneal Neuropathies

ARMS (2):
- FES (Experimental): All subjects will receive a 15-30 minutes a day treatment for 5 days a week. When the subjects achieves the ability to walk with supervision, but with no physical assistance, safely and consistently during the physiotherapy sessions, then either the FES will be provided to the subject to allow ongoing gait practice with the nursing staff in the ward environment. After discharge, the assistive device will be provided for home usage till the end of the research.
  Interventions: Device: FES
- Conventional (No Intervention): Treated with regular gait re-education with or without AFO fitting. All subjects will receive a 15-30 minutes a day treatment for 5 days a week. When the subjects achieves the ability to walk with supervision, but with no physical assistance, safely and consistently during the physiotherapy sessions, then either the AFO will be provided to the subject to allow ongoing gait practice with the nursing staff in the ward environment. After discharge, the assistive device will be provided for home usage till the end of the research.

INTERVENTIONS:
Device: FES
  Other Names: Mygait
  Arms: FES

SUMMARY:
The investigators hypothesize that the gait pattern of following the utilization of a functional electrical stimulation device will be much improved when compared to the effect of regular gait re-education with ankle-foot-orthosis (AFO) fitting in patients in early stages following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute stroke patients suffering a first stroke with clinical presentation, according to the WHO definitions
* Patients suffering from unilateral foot drop
* Independent ambulation before the stroke
* Cognitive and cooperative ability to follow simple instructions
* Neurological condition severity mild to moderate (between 3 and 15, according to the National Institutes of Health Stroke Scale; NIHSS).
* Ability to walk with or without a walking aid (cane, walker), with or without assistance. Functional Ambulation Classification (FAC) of at least 2
* Independently capable to understand an informed consent form.

Exclusion Criteria:

* Cognitive disorders preventing the subject from understanding the trial protocol or following the researcher's instructions
* Orthopaedic injury to the paretic or non-paretic limbs
* Motor disability due to neurological diagnosis, e.g. multiple sclerosis, cerebral palsy, spinal cord injury, and Parkinson
* Peripheral injury of the peroneal nerve or sciatic nerve
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in velocity of gait | Baseline, 4 weeks and 12 week follwing baseline
  Measured in m/s and the change will be in %
Change in step length | Baseline, 4 and 12 weeks following baseline
  Measured in cm and the change will be in %

SECONDARY OUTCOMES:
Gait symmetry | Baseline, 4 and 12 weeks following baseline
  Calculated symmetry of stance duration, swing duration, double support duration, step length, base width, and foot progression
Muscle activity patterns | Baseline, 4 and 12 weeks following baseline
  Surface electromyography (EMG) electrodes will be attached to 6 muscles for evaluation of dynamic muscle activation pattern during gait without the intervention. Specifically, we will monitor the medial gastrocnemius, soleus and tibialis anterior, bilaterally.
Functional assessment | At baseline, 4 and 12 weeks following baseline
  Selective motor control during dorsiflexion will be tested with and without flexed knee according to the classification of three levels: normal, impaired, and unable. This test will be utilized for matching of the test group and control group. Physical evaluation will be conducted to assess the muscle tonus of the gastrocnemius, tibialis anterior and quadriceps according to Ashwart scale. Passive joint range of motion will also be assessed.
  Functional evaluation of each subject will be accomplished using the 10-meter walk. The Functional Ambulation Classification (FAC) will also be applied in order to obtain a patient prognosis level with regard to ambulation.
  Time up and Go (TUG) test will be performed in the in gait laboratory so that the performance of the subjects during the trials can be videotaped.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel